CLINICAL TRIAL: NCT04073303
Title: BOTOX® (onabotulinumtoxinA) Treatment of Masseter Muscle Prominence: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: BOTOX® Treatment for Adults With a Wide Lower Face Due to Masseter Muscle Prominence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1789-301-008
Record Dates: First submitted 2019-08-22; First posted 2019-08-29 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Masseter Muscle Prominence
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Botulinum Toxin Type A (BOTOX®) (Active Comparator): Botulinum Toxin Type A (BOTOX ®) will be administered on Day 1 as bilateral intramuscular injections into the masseter with the possibility of 2 additional treatments
  Interventions: Biological: Botulinum Toxin Type A
- Placebo (Placebo Comparator): Placebo (normal saline) will be administered on Day 1 as bilateral intramuscular injections into the masseter
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Botulinum Toxin Type A — Day 1 Administration of bilateral intramuscular injections into the masseter
  Other Names: OnabotulinumtoxinA; BOTOX®
  Arms: Botulinum Toxin Type A (BOTOX®)
Other: Placebo — Day 1 Administration of bilateral intramuscular injections of placebo (normal saline) into the masseter
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the safety and effectiveness of administering BOTOX for the treatment of Masseter Muscle Prominence (MMP) in adults.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Masseter prominence at the Day 1 visit
* BMI ≤ 30 kg/m2 using the calculation: BMI = weight (kg)/[height (m)]2
* A female participant must be willing to minimize the risk of inducing pregnancy for the duration of the clinical study and follow-up periods

Exclusion Criteria:

* Any medical condition that may put the participant at increased medical risk with exposure to BOTOX, including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other condition that might interfere with neuromuscular function
* An anticipated need for surgery or overnight hospitalization during the study
* An anticipated need for treatment with botulinum toxin of any serotype for any indication during the study (other than study intervention)
* History of dental or surgical procedure for lower facial shaping or masseter muscle reduction
* Prior mid-facial and/or lower facial treatment with nonpermanent soft tissue fillers, synthetic implantations, autologous fat transplantation, fat-reducing injectables, and/or skin-tightening laser treatments within 6 months prior to Day 1
* Prior exposure to botulinum toxin of any serotype to the masseter muscle or lower face at any time, or to any other part of the body within the 6 months prior to Day 1
* History of temporomandibular joint disorder (TMJD)
* Masseter prominence due to other etiologies (eg, parotid gland infection, parotiditis, malignancy)
* Known allergy or sensitivity to any of the components of the study treatments or any materials used in the study procedures
* History of alcohol or drug abuse within 12 months of Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (21):
- Canada (5):
  - Duplicate_Beacon Dermatology Inc /ID# 233018, Calgary, Alberta
  - Duplicate_Humphrey Cosmetic Dermatology /ID# 232764, Vancouver, British Columbia
  - Project Skin MD LTD /ID# 232763, Vancouver, British Columbia
  - Pacific Derm /ID# 233156, Vancouver, British Columbia
  - The Center For Dermatology /ID# 233001, Richmond Hill, Ontario
- China (12):
  - Peking University Third Hospital /ID# 233148, Beijing, Beijing Municipality
  - Duplicate_Peking Union Medical College Hospital /ID# 233072, Beijing, Beijing Municipality
  - Chinese PLA General Hospital /ID# 233158, Beijing, Beijing Municipality
  - Peking University First Hospital /ID# 232973, Xicheng District, Beijing Municipality
  - Tianjin Medical University General Hospital /ID# 232961, Tianjin, Guizhou
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 233008, Wuhan, Hubei
  - Xiangya Hospital Central South University /ID# 233027, Changsha, Hunan
  - Nanjing Drum Tower Hospital /ID# 233016, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University /ID# 232836, Nanjing, Jiangsu
  - Shanghai Ninth People's Hospital,Shanghai Jiaotong University School of Medicine /ID# 232656, Shanghai, Shanghai Municipality
  - Tangdu Hospital of The Fourth Military Medical University, PLA /ID# 233087, Xi’an, Shanxi
  - West China Hospital, Sichuan University /ID# 233107, Chengdu, Sichuan
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 233033, Kaohsiung City, Keelung
  - National Taiwan University Hospital /ID# 233133, Taipei City, Taipei
  - Taipei Medical University Hospital /ID# 233009, Taipei
  - Tri-Service General Hospital /ID# 233080, Taipei

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 377 participants were enrolled and randomized into the study; 284 to BOTOX and 93 to Placebo. A total of 370 participants were included in the modified ITT (mITT) Population; 278 to BOTOX and 92 to Placebo. A participant was considered to have completed the study if he/she had at least completed the treatment visit and the end of study visit.
Pre-assignment Details: The mITT population, consisting of all randomized subjects with at least 1 postbaseline MMPS assessment, comprised 370 subjects.
Groups:
- Placebo: Placebo was administered as bilateral intramuscular injections into the masseter on Day 1.
- BOTOX®: BOTOX ® was administered as bilateral intramuscular injections into the masseter on Day 1, with the possibility of 2 additional treatments
Period: Overall Study
Arm/Group | Placebo | BOTOX®
Started | 93 | 284
mITT Population | 92 | 278
Completed | 70 | 240
Not Completed | 23 | 44
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 16 | 36
Not completed — Lost to Follow-up | 6 | 1
Not completed — Protocol Deviation | 0 | 4
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat (mITT) Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BOTOX® | Total
Number analyzed (Participants) | 92 | 278 | 370
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.0 (8.67) | 31.5 (8.35) | 31.4 (8.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 244 | 326
  Male | 10 | 34 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 91 | 274 | 365
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 76 | 247 | 323
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 0 | 1
  White | 15 | 29 | 44
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Baseline Masseter Muscle Prominence Scale (MMPS) [Count of Participants; unit: Participants] — The investigator assessed the severity of the participant's masseter muscle prominence (MMP) using the MMPS 5-point scale ranging from 1=minimal to 5=very marked. Higher scores represent more severe outcomes.
  Participants
    4 = Marked | 59 | 177 | 236
    5 = Very Marked | 33 | 101 | 134

OUTCOME MEASURES:

1. Primary Outcome: Achievement of ≥ 2-Grade Improvement From Baseline on the Masseter Muscle Prominence Scale (MMPS) at Day 90
Description: Proportion of participants who achieve ≥ 2-grade improvement from baseline at Day 90, per investigator assessments of MMP using the Masseter Muscle Prominence Scale (MMPS).
  MMPS ranges from 1 = minimal to 5 = very marked.
Time Frame: Day 90
Population: mITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BOTOX®
Number analyzed (Participants) | 92 | 278
percentage of participants | 2.2 [0.0 to 5.2] | 51.2 [45.2 to 57.2]
Statistical Analysis 1: Comparison: Placebo vs BOTOX®; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Rate-Difference = 49.0, 95% CI 2-sided [40.1 to 54.1]

2. Secondary Outcome: Achievement of MMPS Grade ≤ 3 at Day 90
Description: Proportion of participants who achieve MMPS Grade of ≤ 3 at Day 90, per investigator assessments of MMP using the Masseter Muscle Prominence Scale (MMPS).
  MMPS ranges from 1 = minimal to 5 = very marked.
Time Frame: Day 90
Population: mITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BOTOX®
Number analyzed (Participants) | 92 | 278
percentage of participants | 9.9 [3.8 to 16.1] | 81.1 [76.4 to 85.9]
Statistical Analysis 1: Comparison: Placebo vs BOTOX®; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Rate-Difference = 71.2, 95% CI 2-sided [60.7 to 76.3]

3. Secondary Outcome: Achievement of MMPS-P Grade ≤ 3 on Day 90
Description: Proportion of participants who achieve MMPS-P Grade ≤ 3 at Day 90, according to participant, per Masseter Muscle Prominence Scale-Participant (MMPS-P)
  MMPS-P ranges from 1 = not at all pronounced to 5 = very pronounced.
Time Frame: Day 90
Population: mITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BOTOX®
Number analyzed (Participants) | 92 | 278
percentage of participants | 19.5 [11.2 to 27.8] | 76.2 [71.1 to 81.4]
Statistical Analysis 1: Comparison: Placebo vs BOTOX®; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Rate-Difference = 56.7, 95% CI 2-sided [45.6 to 64.5]

4. Secondary Outcome: Achievement of MMPS-P ≥ 2-Grade Improvement From Baseline at Day 90
Description: Proportion of participants who achieve ≥ 2-grade improvement from baseline at Day 90, per Masseter Muscle Prominence Scale-Participant (MMPS-P)
  MMPS-P ranges from 1 = not at all pronounced to 5 = very pronounced.
Time Frame: Day 90
Population: mITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BOTOX®
Number analyzed (Participants) | 92 | 278
percentage of participants | 9.1 [3.1 to 15.0] | 58.8 [52.9 to 64.7]
Statistical Analysis 1: Comparison: Placebo vs BOTOX®; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Rate-Difference = 49.7, 95% CI 2-sided [40.6 to 57.4]

5. Secondary Outcome: Achievement of PSAC Grade ≥ 1 (at Least Minimally Improved From Baseline) on Day 90
Description: Proportion of participants who achieve Grade ≥ 1 on Participant Self-Assessment of Change (PSAC) (at least minimally improved from baseline) at Day 90
  PSAC ranges from 3 = much improved to -3 = much worse.
Time Frame: Day 90
Population: mITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | BOTOX®
Number analyzed (Participants) | 92 | 278
percentage of participants | 20.4 [12.0 to 28.7] | 90.8 [87.3 to 94.4]
Statistical Analysis 1: Comparison: Placebo vs BOTOX®; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Rate-Difference = 70.5, 95% CI 2-sided [59.6 to 77.5]

6. Secondary Outcome: Change From Baseline in Lower Facial Width (mm) at Day 90
Description: Calculated from standardized images, measured in millimeters (mm)
Time Frame: Day 90
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: millimeters (mm)
Arm/Group | Placebo | BOTOX®
Number analyzed (Participants) | 92 | 278
millimeters (mm) | -0.04 (0.202) | -5.24 (0.121)
Statistical Analysis 1: Comparison: Placebo vs BOTOX®; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean of Difference = -5.19, 95% CI 2-sided [-5.64 to -4.75]

7. Secondary Outcome: Median Duration of Effect for MMPS Responders
Description: Median duration of effect for BOTOX-treated MMPS responders.
Time Frame: Up to Day 360
Population: mITT Population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | BOTOX®
Number analyzed (Participants) | 278
Days
  MMPS ≥ 2-Grade Improvement: number analyzed (Participants) | 133
  MMPS ≥ 2-Grade Improvement | 176.0 [154.0 to 183.0]
  MMPS Grade ≤ 3: number analyzed (Participants) | 208
  MMPS Grade ≤ 3 | 213.0 [204.0 to 236.0]
  MMPS ≥ 1-Grade Improvement: number analyzed (Participants) | 231
  MMPS ≥ 1-Grade Improvement | 268.0 [239.0 to 304.0]

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from the start of safety data collection/time of informed consent/enrollment (whichever study team prefers per protocol/study design) to the end of the study. The median time on follow-up (or mean time followed) was 539.0 and 540.0 Days for Placebo and BOTOX ®, respectively.
Arm/Group | Placebo | BOTOX®
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/283
Serious Adverse Events (participants affected / at risk) | 4/93 | 11/283
Other Adverse Events (participants affected / at risk) | 19/93 | 54/283
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=93) | BOTOX® (N=283)
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 (0) | 1 (1)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GALLBLADDER POLYP (Hepatobiliary disorders) | 0 (0) | 1 (1)
POST-ACUTE COVID-19 SYNDROME (Infections and infestations) | 0 (0) | 1 (1)
PULMONARY TUBERCULOSIS (Infections and infestations) | 0 (0) | 1 (1)
POST HERPETIC NEURALGIA (Nervous system disorders) | 1 (1) | 0 (0)
ABORTION OF ECTOPIC PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
ABORTION THREATENED (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
FOETAL GROWTH RESTRICTION (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
ENDOMETRIOSIS (Reproductive system and breast disorders) | 1 (1) | 0 (0)
FALLOPIAN TUBE CYST (Reproductive system and breast disorders) | 0 (0) | 1 (1)
LUNG OPACITY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
NASAL SEPTUM DEVIATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ABORTION INDUCED (Surgical and medical procedures) | 1 (1) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=93) | BOTOX® (N=283)
NASOPHARYNGITIS (Infections and infestations) | 3 (4) | 17 (19)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 6 (7) | 18 (22)
MASTICATION DISORDER (Musculoskeletal and connective tissue disorders) | 6 (6) | 14 (17)
HEADACHE (Nervous system disorders) | 6 (8) | 11 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT04073303/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/03/NCT04073303/SAP_001.pdf